CLINICAL TRIAL: NCT05798325
Title: Feasibility, Validation and Application of Digital Tools for the Follow-up of Neuromuscular Patient
Brief Title: Feasibility, Validation and Application of Digital Tools for the Follow-up of Neuromuscular Patient Mobility in Daily Living
Acronym: DT4RD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Myologie, France (Other)
Collaborators: Aparito Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DT4RD
Record Dates: First submitted 2023-03-08; First posted 2023-04-04 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular Diseases; Dystrophy; Monitoring; Accelerometer; Evaluation
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Spirometry; Arthrometry, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Principal (Other)
  Interventions: Other: 2MWT; Other: MFM32; Other: MyoGrip; Other: QOL-gNMD; Diagnostic Test: Spirometry; Device: Acceleromerty; Other: 10mWT; Other: PUL; Other: NSAA; Other: NSAD; Other: TANS; Other: MyoPinch; Other: MyoQuad; Other: ACTIVLIM; Other: PREM; Other: SF-MPQ; Other: FSS; Other: IPAQ; Other: Rang of motion; Device: Goniometry; Other: Video captured monitoring; Device: Activity monitoring

INTERVENTIONS:
Other: 2MWT — Two minutes walk tests.
  Other Names: Two minutes walk tests
Other: MFM32 — Motor Function Measurement (MFM) is a quantitative scale created to measure global motor functional abilities in a person with neuromuscular disease.
  Other Names: Muscle Motor Function 32
Other: MyoGrip — The MyoGrip is a dynamometer for measuring grip strength.
Other: QOL-gNMD — The "Quality of Life in genetic Neuromuscular Disease" questionnaire (QoL-gNMD) is a patient reported outcome measure (PROM) tool specifically designed for patients with a lowly progressive neuromuscular disease with genetically predominant muscular damage
Diagnostic Test: Spirometry — Forced vital capacity (FVC), peak expiratory flow (PEF) and forced expiratory volume in 1 second (FEV1) will be measured in the hospital with the local hospital device (e.g. Vitalograph) under the supervision of the clinical evaluator, and at home with a portable device.
  Other Names: Spirobank Smart
Device: Acceleromerty — The Links sensor system is a measuring device and consists of the Links Pods and the Links Hub. The Links pods contain an accelerometer, gyroscope and magnetometer to measure position relative to a global reference frame.
  Other Names: Links sensor system
Other: 10mWT — 10 meters walking Test.
Other: PUL — The Performance of the Upper Limb (PUL) is a functional scale specifically designed for assessing upper limb function in Duchenne muscular dystrophy.
  Other Names: Performance of Upper Limb
Other: NSAA — The North Star Ambulatory Assessment (NSAA) is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy.
  Other Names: North Star Ambulatory Assessment
Other: NSAD — The NSAD was developed to measure motor performance in ambulant and non-ambulant subjects as part of the clinical outcome study of dysferlinopathy.
  Other Names: North Star Assessment for limb-girdle type muscular dystrophies
Other: TANS — This scale is derived from the North Star Ambulatory Assessment and several items from the Egan Klassifikation Scale (EK2).
  Other Names: Transition Assessment North Star
Other: MyoPinch — The MyoPinch is a high-precision dynamometer that allows the evaluation of key pinch strength.
Other: MyoQuad — The MyoQuad is a high-precision dynamometer that allows the evaluation of knee extension strength.
Other: ACTIVLIM — Activity limitations, as measured by ACTIVLIM, is defined as the difficulties a patient may have in executing daily activities, whatever the strategies involved.
Other: PREM — This questionnaire is made up of simple questions relating to the assessments and assessment tools that were used during the study.
  Other Names: Patient Reported Experience Measures
Other: SF-MPQ — The main component of the SF-MPQ consists of 15 descriptors (11 sensories; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  Other Names: Modified Short-form McGill Pain Questionnaire
Other: FSS — The Fatigue Severity Scale is used to assess the severity of fatigue and its impact on daily living. The patient responds on a Likert-type scale ranging from 1 to 7.
  Other Names: Fatigue Severity Scale
Other: IPAQ — This questionnaire assesses overall physical activity and the level of sedentary lifestyle during the last seven days.
  Other Names: International Physical Activity Questionnaire
Other: Rang of motion — The EasyAngle® is a digital goniometer improving long established goniometric functionality with rotation, inclination, and scoliosis measurement capabilities.
  Other Names: EasyAngle
Device: Goniometry — The Links sensor system is a measuring device and consists of the Links Pods and the Links Hub. The Links pods contain an accelerometer, gyroscope and magnetometer to measure position relative to a global reference frame.
  Other Names: Links Sensor System goniometers
Other: Video captured monitoring — Once every four weeks, while wearing the Yumen electronic goniometers (Links Sensor System), the patients will be asked to record on video three tasks related to:
  1. Upper limbs: hands to head
  2. Lower limbs: Sit to stand with or without the help of a person
  3. Self-defined important task: A task of the patient's choice, from a list of tasks, representative of his/her motor difficulties or hindrance to autonomy.
Device: Activity monitoring — Wearable devices (connected watch) will collect health-related data on a 24/7 basis remotely as patients go through their daily routines at home and work.
  Other Names: Activity assessment and physiological parameters

SUMMARY:
The low prevalence of rare diseases hinders the design of clinical studies with sufficient statistical power to demonstrate the efficacy of new drugs. This can only be achieved by setting up international multicentre studies, which is challenging due to a lack of objective, universal outcome measures that generate high-quality, reproducible data. One of the hurdles in attaining universal outcome measures for clinical trials is the difficulty to capture and distinguish ambulatory from non-ambulatory, autonomous and assistive or involuntary movements. This makes a trial assessing the ambulatory phase very challenging at this moment. Excluding many participants from trials and many patients from access to medication.

Integration and validation of the technology in trials, research and patients' lives is essential in overcoming this hurdle. For example, in dystrophinopathies separate outcome measures exist for ambulant and non-ambulant participants, but the relation between these outcome measures or a transitional outcome measure/end point is largely missing.

Following an exhaustive literature review, several tools have been selected to remotely follow various symptoms of neuromuscular patients including weakness, pain, fatigue, cognitive defects, motor impairments (including loss of dexterity, ataxia...), metabolic, respiratory and cardiac troubles, contractures, tremor, falls, hypo or hypersomnia... The toolbox includes common measures for all patients but may include additional measures specific to the patient's symptoms (hence in turn to the patients' disease).

The measurements are designed to not be invasive, intrusive or burdensome for the patient.

DT4RD is going to leverage state-of-the art technology, clinical rating scales and psychometric/data analysis to deliver fit for purpose remote clinical assessments of mobility to ensure maximum patient benefit, specifically:

* Compare face to face clinical data collected in hospital with Patient Generated Data recorded remotely
* Examine how sensors can enhance measurement potentially at home and during clinical visits
* Promote a clear focus on user centered design and the integration of technology
* Use reliability and validity analyses to equate any common measures (those with the same or a similar construct)
* Demonstrate a proof-of-concept model into which different measures can be interchangeable

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 60 years
* Patients with a genetically confirmed/molecular-proven neuromuscular or neurometabolic disease*
* Patients experiencing walking difficulties in the home and at high risk of limiting participation and walking outside of the home.
* Written informed consent
* Able to comply with all protocol requirements, including video recording
* Affiliated to or beneficiary of a social security scheme (for France)

Exclusion Criteria:

* Patients with undefined diagnosis or any diagnosis other than neuromuscular or neurometabolic disease
* Patient walking 10m in less than 10s
* Guardianship/trusteeship
* Pregnant or nursing women
* Patients having relevant concomitant pathologies that, in the appreciation of the investigator could interfere with protocol compliance
* Patients not being affiliated with local social security (for France)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Global home evaluations' attendance | Through study completion, an average of 1 year
  Proportion of home assessments carried out compared to the number of home assessments planned

SECONDARY OUTCOMES:
Compliance with filling out questionnaires at home | Through study completion, an average of 1 year
  Analysis of the proportion of replies to the questionnaires at home
Compliance regarding using of the spirometer at home | Through study completion, an average of 1 year
  Analysis of the proportion of valid spirometry data collected at home
Compliance regarding using of the LINKS sensors device at home | Through study completion, an average of 1 year
  Analysis of the proportion of usable accelerometry data collected at home
Compliance regarding using of the activity sensor at home | Through study completion, an average of 1 year
  Analysis of the proportion of usable data collected at home using the smartwatch
Compliance regarding achievement of video tasks at home | Through study completion, an average of 1 year
  Analysis of the usability of the video tasks performed at home
Correlation of home and hospital spirometer Forced vital capacity measurements | Through study completion, an average of 1 year
  Comparison of Forced vital capacity data collected during home and hospital spirometer measurements
Correlation of home and hospital spirometer peak expiratory flow measurements | Through study completion, an average of 1 year
  Comparison of Peak expiratory flow data collected during home and hospital spirometer measurements
Correlation of home and hospital spirometer forced expiratory volume in 1 second measurements | Through study completion, an average of 1 year
  Comparison of forced expiratory volume in 1 second data collected during home and hospital spirometer measurements

CONTACTS AND LOCATIONS:
Locations (2):
- Association Institut de Myologie, Paris, France
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided